CLINICAL TRIAL: NCT01228201
Title: Physical Exercise and Coronary Artery Plaque Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trondheim University Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Rune Wiseth, Professor Rune Wiseth, Trondheim University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTNU - project no 46028000
Record Dates: First submitted 2010-10-21; First posted 2010-10-26 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerboic interval training (Experimental)
  Interventions: Behavioral: Aerobic interval training
- Moderate continuous training (Active Comparator)
  Interventions: Behavioral: Moderate continuous training

INTERVENTIONS:
Behavioral: Moderate continuous training — Three training sessions per week in a total of 12 weeks
  Arms: Moderate continuous training
Behavioral: Aerobic interval training — Three training sessions per week in a total of 12 weeks
  Arms: Aerboic interval training

SUMMARY:
The purpose of this study is to examine the effect of two different physical exercise protocols on changes in coronary artery plaque composition and development of in-stent restenosis in patients treated with percutaneous coronary intervention with stent implantation. The investigators will compare aerobic interval training and moderate continuous training. Both exercise protocols have a duration of 12 weeks. The investigators hypothesize that aerobic interval training is superior to moderate continuous training regarding effects on the composition of coronary artery plaques and a reduction in the development of in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* stable or unstable coronary artery disease treated with percutaneous coronary intervention with stent implantation,
* informed patient consent

Exclusion Criteria:

* ST-elevation myocardial infarction,
* inability to give informed consent,
* inability to participate in regular training due to residency, work situation or comorbidity,
* any known chronic inflammatory disease other than atherosclerosis,
* planned surgery within the next four months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Artery plaque composition evaluated by intravascular ultrasound and virtual histology | After 12 weeks
  Findings at 12 weeks will be compared to baseline results

SECONDARY OUTCOMES:
Occurrence of in-stent restenosis related to endothelial dysfunction, inflammatory biomarkers and the dimension of the main left coronary artery | After 12 weeks
  Findings at 12 weeks will be compared to baseline results

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, M.D, PhD, Principal Investigator — Department of Cardiology, Trondheim University Hospital
Locations (1):
- Department of Cardiology, Trondheim, Norway

REFERENCES:
- [Background] Munk PS, Staal EM, Butt N, Isaksen K, Larsen AI. High-intensity interval training may reduce in-stent restenosis following percutaneous coronary intervention with stent implantation A randomized controlled trial evaluating the relationship to endothelial function and inflammation. Am Heart J. 2009 Nov;158(5):734-41. doi: 10.1016/j.ahj.2009.08.021. PMID 19853690
- [Derived] Taraldsen MD, Wiseth R, Videm V, Bye A, Madssen E. Associations between circulating microRNAs and coronary plaque characteristics: potential impact from physical exercise. Physiol Genomics. 2022 Apr 1;54(4):129-140. doi: 10.1152/physiolgenomics.00071.2021. Epub 2022 Feb 28. PMID 35226566